CLINICAL TRIAL: NCT00861315
Title: Phase II Study of High Dose Nebulized Amikacin in Patients With Pneumonia Undergoing Mechanical Ventilation
Brief Title: Pharmacokinetics of Nebulized Amikacin in Patients With Pneumonia Undergoing Mechanical Ventilation
Acronym: DARTAGNAN
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Pour La Promotion A Tours De La Reanimation Medicale (Other)
Responsible Party: Pr Dominique Perrotin, Association Pour La Promotion A Tours De La Reanimation Medicale
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DARTAGNAN
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Pneumonia; Nebulization; Amikacin
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nebulized amikacin (Experimental): Patients receive nebulized amikacin once a day during three days. Placebo is administered intravenousely
  Interventions: Drug: Nebulized amikacin; Drug: Placebo infusion
- Intravenous amikacin (Active Comparator)
  Interventions: Drug: Intravenous amikacin; Drug: Placebo nebulization

INTERVENTIONS:
Drug: Nebulized amikacin — Amikacin is nebulized at a dose of 60 mg/Kg (6 first patients of the arm), 80 mg/Kg (6 subsequent patients) or 100 mg/Kg (last 6 patients of the arm)
  Arms: Nebulized amikacin
Drug: Intravenous amikacin — 20 mg/Kg amikacin are administred intravenousely once a day during three days.
  Arms: Intravenous amikacin
Drug: Placebo nebulization — 0.9% saline solution is nebulized once a day during three days
  Arms: Intravenous amikacin
Drug: Placebo infusion — 0.9% saline is administered intravenousely once a day during three days
  Arms: Nebulized amikacin

SUMMARY:
Inclusion of patients undergoing mechanical ventilation and presenting a pneumonia in order to determine serum pharmacokinetics of nebulized amikacin. The primary aim is to determine the dose of amikacin to be nebulized in order to observe amikacin serum concentrations close to but inferior to those observed after standart intravenous amikacin infusion.

DETAILED DESCRIPTION:
After inclusion, patients undergo intravenous infusion of 20 mg/Kg of amikacin with amikacin serum concentrations being monitored over the following 24 hours.

Randomization occures after this first amikacin infusion. Patients are randomized to group nebulized amikacin or intravenous amikacin. The three next days of the study patients recieve nebulized amikacin (or nebulized placebo) during mechanical ventilation and a placebo infusion (amikacin infusion in case of placebo nebulization) using a air driven jet nebulizer. Amikacin serum concentrations are monitored over 24 hours after each nebulization.

Patients are followed up during 10 days for safety and efficacy. The dose of amikacin to be nebulized is 60 mg/Kg for the first 6 patients (phase A), 80 mg/Kg for the next 6 patients (phase B) and 100 mg/Kg for the last 6 patients (phase C). Each phase is started after review of the results of the preceeding phase by an idependent safety and monitoring board.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to intensive care unit.
* Patients undergoing mechanical ventilation for more than 48H.
* Suspicion of ventilator associated pneumonia.

Exclusion Criteria:

* Allergy to amikacin or any compound of the medication.
* Body mass index > 30 kg/m2.
* Myasthenia gravis.
* Acute or chronic renal failure.
* Vestibulo-cochlear disease.
* Pregnancy.
* Brain death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Determintion of nebulized amikacin dose (60 mg/Kg, 80 mg/Kg or 100 mg/Kg) which results in serum amikacin concentrations equal or below the serum amikacin concentrations measured after 20 mg/Kg intravenous amikacin infusion

SECONDARY OUTCOMES:
Comparison of clinical pulmonary infection score evolution between patients treated with nebulized amikacin and patients treated with intravenous amikacin | 10 days
Comparison of serum procalcitonin concentration evolution between patients treated with nebulized amikacin and patients treated with intravenous amikacin | 10 days
Comparison of c reactive protein evolution between patients treated with nebulized amikacin and patients treated with intravenous amikacin | 10 days
Comparison duration of mechanical ventilation between patients treated with nebulized amikacin and patients treated with intravenous amikacin | 10 days

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service de réanimation médicale polyvalente. Hôpital Bretonneau CHRU, Tours, Indre et Loire
  - Service de réanimation médicale. Hôpital La Source. CH Orléans, Orléans, Loiret